CLINICAL TRIAL: NCT04986280
Title: Diagnostic Accuracy and Performance of 18F-PSMA-1007 in the Detection of Recurrent Prostate Cancer - a Prospective, Single-arm Study
Brief Title: Diagnostic Accuracy and Performance of 18F-PSMA-1007
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01383
Record Dates: First submitted 2021-04-12; First posted 2021-08-02 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
Keywords: PSMA; Recurrent prostate cancer; Diagnostic accuracy; 18F-PSMA-1007; [18F]PSMA-1007
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Arm 1 - All patients will undergo PET/CT with 18F-PSMA-1007
  Interventions: Diagnostic Test: [18F]PSMA-1007

INTERVENTIONS:
Diagnostic Test: [18F]PSMA-1007 — PSMA PET/CT using the intervention.
  Other Names: F-18-PSMA-1007

SUMMARY:
Whereas 18F-PSMA-1007 has rapidly established itself as a radiotracer for the investigation of prostate cancer, there are no studies confirming its diagnostic performance. The purpose of this study is to determine the diagnostic performance for this radiotracer.

DETAILED DESCRIPTION:
In this prospective, single-armed diagnostic imaging study men undergoing standard-of-care PSMA PET/CT using [18F]PSMA-1007 shall be studied. The primary objective is to confirm the positive predictive value (PPV) of this tracer at a patient-based level by recruiting until 53 patients with follow-up to a composite reference standard are available. Secondary outcomes shall include patient based rate of pathological-scans stratified by PSA, the PPV stratified by region , interrelate agreement, frequency of indeterminate lesions and the safety and tolerability of the examination.

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients referred for investigation of recurrent PC by PSMA PET/CT.
* Patients with known biochemical recurrence of a histologically confirmed primary prostate cancer, defined as:

Post prostatectomy: two consecutive PSA > 0.2 ng/ml Post-radiotherapy: a rise of 2ng/mL > post-therapy nadir (ASTRO consensus definition)

* Male patients >18 years old
* PSA measured ± 4 weeks of the PSMA-PET/CT
* Patients willing and able to consent to the informed consent document

Exclusion Criteria:

* Patients with ADT within 6 months prior to the PSMA-PET/CT
* Inability to provide informed, written consent
* Patients undergoing active treatment for a second non-prostatic malignancy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data will be obtained prospectively from patients referred for routine 18F-PSMA-11 PET/CT for recurrent prostate cancer at the university clinic for nuclear medicine, Inselspital Bern. Follow up data (further imaging, laboratory parameters and details of further treatment) will be collected up to 12 months' follow up from the date of examination.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Primary objective: To confirm the PPV of the new tracer (patient-based PPV) | At one year follow up
  The primary end point is the per patient PPV for the detection of PSMA-positive tumour lesions as confirmed by either a) histology or b) a composite reference standard of imaging and/or PSA fall following focal therapy in the absence of systemic therapy.

SECONDARY OUTCOMES:
• To determine the patient-based detection rate of pathologic scans (sensitivity) for the new tracer | Within one week of scan
  Patient based detection (PET-positivity) rate (stratified by PSA value)
To explore the regional based PPV | At one year follow up
  Region-based PPV (prostate bed, pelvic lymph nodes, extra-pelvic lymph nodes, extra-pelvic viscera and bone metastases)

OTHER OUTCOMES:
To calculate the inter-reader reliability | Within one month of scan
  The interrater agreement (ordinal scale, no units) for PET-findings will be determined. The joint-interrate reliability will be compared by a combined assessment of Fleiss' kappa and Krippendorf's alpha.
Frequency of diagnostic pitfalls or indeterminate lesions requiring follow-up | Within one month of scan
  The frequency of indeterminate lesions requiring follow up / indeterminate lesions will be recorded by all readers and analysed by descriptive statistics
Number of patients with adverse events. | Up to 48 hours follow up post scan
  Patients will be contacted by phone one to three days post imaging and assessed for adverse events (AE). Any reported events will be followed up by a physician in the clinic for study related adverse events requiring further evaluation. Adverse events are as defined in supplementary materials and will be recorded using the AE form in the eCRF.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Afshar-Oromieh, MD, Study Chair — Deputy Clinic Director
Locations (1):
- Inselspital, Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request